CLINICAL TRIAL: NCT05102513
Title: Unilateral Cleft Lip Closure - Development of a New Hybrid Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marco Kesting (Other)
Responsible Party: Sponsor-Investigator, Marco Kesting, Prof. Dr. med. Dr. med. dent., University Hospital Erlangen
Organization: University Hospital Erlangen (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20211010
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Complete Unilateral Cleft Lip
Keywords: Cleft Lip; Cleft Lip Repair; Unilateral Cleft Lip
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: 20 complete unilateral cleft lips are operated; 10 are treated with the Millard II technique and 10 are treated with the new hybrid technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Cleft Lip Repair with the New Hybrid Technique (Experimental)
  Interventions: Procedure: Unilateral Cleft Lip Repair: Hybrid Technique
- Unilateral Cleft Lip Repair with the Millard II Technique (Active Comparator)
  Interventions: Procedure: Unilateral Cleft Lip Repair: Millard 2 Technique

INTERVENTIONS:
Procedure: Unilateral Cleft Lip Repair: Hybrid Technique — The rotation flap of the Millard II technique was expanded by extending the incision into the columella - similar to the well-known Mohler technique. The caudal part of the advancement flap of the Millard II technique was lengthened by a wave cut as known from the Pfeiffer procedure. For the vermillion a Noordhoff plasty is applied.
  Arms: Unilateral Cleft Lip Repair with the New Hybrid Technique
Procedure: Unilateral Cleft Lip Repair: Millard 2 Technique — A curved incision is marked skirting the philtral ridge. If more length is required a back-cut incision can be performed. The C-flap is outlined by the incision just marked and the incision along red-white border up to the base of the columella. On the cleft side an advancement flap is designed. For the vermillion a Noordhoff plasty is applied.
  Arms: Unilateral Cleft Lip Repair with the Millard II Technique

SUMMARY:
Unilateral cleft lips can be treated with different incision techniques. According to a survey by the American Cleft Palate Association, the Millard II technique is currently used by the majority of US cleft surgeons. In this technique, a cleft-sided advancement flap is pivoted from the cleft side into the rotation flap of the non-cleft side, which serves, among other things, to lengthen the lip. However, the rotational component is often insufficient to sufficiently lengthen the lip on the cleft side. The result is a raised red lip, a shortened edge of the philtrum or a so-called pipe-hole deformity. In order to compensate for these "deficiencies", a triangular flap is currently being formed in the area of the white roll, which is intended to provide sufficient lengthening.

However, the scar of the triangular flaps runs exactly opposite to the aesthetic unit. In addition, it often provides a step formation within the white roll. Knowing the weaknesses of the previous techniques, a further development of the incision was made. The rotational flap of the Millard II technique was extended by extending the incision into the columella - similar to the well-known Mohler technique. The caudal part of the advancement flap of the Millard II technique was extended by a wave incision as known from the Pfeifer procedure.

ELIGIBILITY:
Inclusion Criteria:

* Complete unilateral cleft lip and palate

Exclusion Criteria:

-

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the length of the philtral colomn on the cleft and non-cleft side | perioperatively to 6 month postoperatively
  Perioperatively, a 3-D scan and photos are taken. Additional photos are also taken after the removal of the stitches, after 3 months and after 6 months. From these, the increase in length of the philtral column can be determined with 3D computer software and with a linear measurement of the photos.
Angle of the columella | perioperatively
  A 3d scan and photos are made perioperatively. From this the angle of the columella can be determined with a 3D Computer software and with a linear measurement of the photos.
Distance from the midpoint of the columella to the lateral alae | perioperatively
  Perioperatively, a 3-D scan and photos are taken. The distance can be measured with a 3D computer software and with a linear measurement of the photos.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Kesting, Prof Dr Dr, Principal Investigator — Mund-, Kiefer- und Gesichtschirurgie Erlangen
Locations (1):
- Mund-, Kiefer- und Gesichtschirurgische Klinik, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No